CLINICAL TRIAL: NCT00055068
Title: Family Based Treatment of Early Childhood OCD
Brief Title: Family Based Treatment of Early Childhood Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH060669 (NIH); R21MH060669 (NIH); DSIR CT-S
Record Dates: First submitted 2003-02-19; First posted 2003-02-20 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2008-02

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Relaxation Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT)
Behavioral: Relaxation Training

SUMMARY:
This study will evaluate a treatment program for young children with Obsessive Compulsive Disorder (OCD) and their families.

DETAILED DESCRIPTION:
Childhood onset OCD is a serious condition that may be a predictor of illness in adulthood. To date, no OCD psychotherapy trials have specifically focused on early childhood. Development of interventions for childhood onset OCD that address both developmental considerations and familial relationships is necessary.

Participants are randomly assigned to receive 12 sessions of either Cognitive Behavioral Therapy (CBT) or Relaxation Training (RT) over the course of 14 weeks. The CBT treatment is designed to lessen anxiety by addressing specific OCD symptoms. The relaxation intervention addresses generalized feelings of anxiety with the expectation that OCD symptoms may benefit indirectly. The clarity, completeness, acceptability, and feasibility of both interventions is assessed. A 3-month post-treatment follow-up is also conducted.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive Compulsive Disorder (OCD)

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2002-03; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital/Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Freeman JB, Garcia AM, Coyne L, Ale C, Przeworski A, Himle M, Compton S, Leonard HL. Early childhood OCD: preliminary findings from a family-based cognitive-behavioral approach. J Am Acad Child Adolesc Psychiatry. 2008 May;47(5):593-602. doi: 10.1097/CHI.0b013e31816765f9. PMID 18356758